CLINICAL TRIAL: NCT00595530
Title: Use of Low-Dose Ketamine Infusion in Acute Painful Episodes of Sickle Cell Disease: A Pilot Study
Brief Title: Low-Dose Ketamine Infusion for Children With Sickle Cell Disease-Related Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment and patient interest in study
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, William Zempsky, MD, Director, Pain Relief Program, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-101
Record Dates: First submitted 2007-12-27; First posted 2008-01-16 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Sickle Cell Disease
Keywords: ketamine; vasoocclusive pain
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): This group will receive ketamine
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — Medication administered via IV. This study will utilize 4 doses of ketamine: 0.05 mg/kg/hr, 0.1 mg/kg/hr, 0.15 mg/kg/hr, and 0.2 mg/kg/hr.
  Dosing Regimen:
  * Patients begin the ketamine infusion at 0.05 mg/kg/hr.
  * 4 or more hrs after infusion is started, the dose may be increased to 0.1 mg/kg/hr if:
    1. patient's pain has not improved to an acceptable level
    2. side effects remain acceptable
  * 4 hrs or more after the previous increase, the dose may be adjusted to 0.15 mg/kg/hr
  * 4 hrs or more after the previous increase, the dose may be adjusted to 0.2 mg/kg/hour
  * Maximum dose of ketamine is limited to 300 mg per 24 hrs
  Patient may receive ketamine up to 72 hrs after initiation.
  Other Names: Ketalar

SUMMARY:
Acute pain episodes associated with sickle cell disease (SCD) are very difficult to manage effectively. Opioid tolerance and side effects have been major roadblocks in our ability to provide these patients with adequate pain relief. This pilot study is designed to examine the safety and feasibility of using ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, in the inpatient seeing with children and adolescents who have sickle cell vasoocclusive pain. Previous research suggests that in subanesthetic doses, ketamine may be able to prevent the development of opiate tolerance and facilitate better pain relief with lower opiate doses, allowing for less respiratory depression, less sedation, easier ambulation, less deconditioning, shorter hospital stays, and better quality of life. The goal of this pilot study is to evaluate the safety and feasibility of using a continuous infusion of ketamine, in conjunction with opiates, in the inpatient setting for sickle cell vasoocclusive pain. It is hypothesized that using a low dose ketamine infusion in conjunction with opiates will be a safe and feasible practice for the treatment of sickle cell pain.

DETAILED DESCRIPTION:
3.2 Study Design/Type

1. Patient meeting inclusion/exclusion criteria is enrolled up to 24 hours after admission for a vasoocclusive episode.
2. Prior to onset of ketamine infusion, the following information is collected:

   1. Demographic information (age, gender, SCD genotype, past history of SCD-related complications) [Obtained from the patient's medical chart]
   2. Opiate utilization/hour since admission [Obtained from the patient's medical chart]
   3. Numerical Rating Scale (NRS) scores since admission [Obtained from the patient's medical chart]
   4. Sedation score (University of Michigan Sedation Scale) is obtained [By the nursing staff]
   5. Body outline figure of the Adolescent Pediatric Pain Tool (validated down to age 7) is administered [By the research staff]
   6. Ketamine Effects Scale (KES) is administered to the patient [By the research staff]
3. Ketamine infusion is begun at 0.05 mg/kg/hour.
4. After infusion is initiated:

   1. Vital signs are taken every hour for two hours after infusion begins, then after two hours, then every four hours for the remainder of the hospitalization [Completed by the nursing staff]
   2. Pain scores are recorded with vital signs if the patient is awake [Completed by nursing staff]
   3. Patient is also asked if pain is a lot better, a little better, no change, a little worse, or a lot worse than previous assessment [Completed by nursing staff]
   4. Sedation score (University of Michigan Sedation Scale) assessed with pain score [Completed by the nursing staff]
   5. Adolescent Pediatric Pain Tool (APPT) body outline figure is completed by the patient once per day between 3 pm and 5 pm. [Administered by the research staff]
   6. Ketamine Effects Scale (KES) is administered to the patient once per day between 3pm and 5pm [By the research staff]
   7. Patient is monitored for side effects including dreams, disorientation, dysphoria, agitation, CNS depression, respiratory depression, increasing hypoxia, nausea, or vomiting [Completed by the nursing or research staff]
   8. Need for supplemental oxygen is recorded (oxygen saturation <95%) [Completed by nursing staff]
   9. Opiate use and NSAID use/6 hours is recorded [Completed by the nursing or research staff]
5. The infusion may be discontinued or decreased at any time due to unacceptable side effects as determined by the clinician, patient, parent, or principal investigator.
6. Agents designed to reduce ketamine side effects [midazolam (Versed), clonidine, lorazepam (Ativan), or diazepam (Valium)] may be administered at the discretion of the attending physician or the principal investigator.
7. 4 hours or more after infusion begins, the infusion rate may be increased to 0.1 mg/kg/hour if the following parameters are met:

   1. patient's pain has not improved to an acceptable range (pain score is still ≥5)
   2. side effects remain acceptable
8. 4 hours or more after the previous increase the ketamine infusion may be increased to 0.15 mg/kg/hour per parameters.
9. 4 hours of more after the previous increase the ketamine infusion may be increased to 0.2 mg/kg/hour per parameters.
10. The ketamine infusion will be discontinued at the time of transition to oral pain medication, or no more than 72 hours after initiation, or at the request of the clinician, patient, parent, or principal investigator.
11. Pain scores, vital signs, sedation score, opiate use, APPT body outline figure, and KES score will be recorded as above for the remainder of the hospitalization.
12. Total length of hospitalization will be recorded.
13. Patient will be contacted on a weekly basis for 4 weeks following hospitalization for review of potential side effects, pain episodes, or events leading to re-admission.
14. The patient's medical record will be reviewed to determine duration of previous hospitalizations for SCD pain in the previous 24 months and opiate utilization, pain scores, and transition to oral opiates during those hospitalizations.

3.3 Randomization

This will be conducted as a pilot study; patients will not be randomized.

3.4 Duration

The length of the patient's participation in this study is the duration of their hospitalization, as well as 4 weeks worth of follow-up phone calls.

3.5 Discontinuation

Individual patients will stop receiving ketamine if they develop acute chest syndrome (ACS), have a stroke, are transferred to the Intensive Care Unit (ICU), if their hemoglobin falls below 5 mg/dl, if they experience unacceptable side effects, or at the request of the PI, attending, patient, or parent. However, they will continue to be in the study and all data will be collected throughout the duration of their hospitalization.

The entire trial will be terminated when 20 patients have completed the protocol, or if there is an unexpected rate of acute chest syndrome or admissions to the pediatric intensive care unit (PICU).

ELIGIBILITY:
Inclusion Criteria:

* CCMC: Children ages 7-22 years (inclusive) with documented sickle cell disease
* UCHC: Adults 18 years (inclusive) and above with documented sickle cell disease
* Sudden onset of acute pain consistent with a vasoocclusive episode -Pain requiring hospitalization, placement on pain protocol, and patient- controlled opiates
* Pain score of greater than or equal to 5 out of 10 when ketamine infusion is started
* Cognitive ability to report pain on a 0 to 10 Numerical Rating Scale (NRS)
* At least one prior hospitalization for vasoocclusive pain at CCMC in the previous 24 months
* Parental consent and child assent

Exclusion Criteria:

* Children hospitalized for a primary diagnosis other than vasoocclusive episode
* Concurrent Acute Chest Syndrome (ACS)
* Hemoglobin < 5 mg/dL
* Concurrent history of glaucoma or raised intracranial pressure
* Signs or symptoms consistent with stroke
* History of liver or renal dysfunction
* Pregnancy (females age 12 and above must have pregnancy test)
* Simultaneous participation in investigational drug study
* Primary language spoken other than English
* No hospitalizations to CCMC for vasoocclusive pain in the previous 24 months

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-03-04 (Actual); Primary Completion 2010-02-12 (Actual); Study Completion 2010-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Zempsky, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data as the low enrollment makes the results of this study non-generalizable.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were recruited from the sickle cell population from PI's clinic and the hematology/oncology clinic
Pre-assignment Details: There were no pre-assignment details
Groups:
- Procedure for Administering Ketamine to SCDpatients: This group will receive ketamine
  ketamine: The medication will be administered intravenously. This study will utilize 4 doses of ketamine: 0.05 mg/kg/hour, 0.1 mg/kg/hour, 0.15 mg/kg/hour, and 0.2 mg/kg/hour.
  Dosing Regimen:
  * All patients will begin the ketamine infusion at 0.05 mg/kg/hour.
  * 4 or more hours after the infusion is started, the dose may be increased to 0.1 mg/kg/hour if:
    1. the patient's pain has not improved to an acceptable level (pain score is still ≥5)
    2. side effects remain acceptable
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.15 mg/kg/hour
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.2 mg/kg/hour
  * The maximum dose of ketamine will be limited to 300 mg per 24 hours
  The patient may receive ketamine up to 72 hours after initiation.
Period: Overall Study
Arm/Group | Procedure for Administering Ketamine to SCDpatients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Protocol for Administering Ketamine to Patients: This group will receive ketamine
  ketamine: The medication will be administered intravenously. This study will utilize 4 doses of ketamine: 0.05 mg/kg/hour, 0.1 mg/kg/hour, 0.15 mg/kg/hour, and 0.2 mg/kg/hour.
  Dosing Regimen:
  * All patients will begin the ketamine infusion at 0.05 mg/kg/hour.
  * 4 or more hours after the infusion is started, the dose may be increased to 0.1 mg/kg/hour if:
    1. the patient's pain has not improved to an acceptable level (pain score is still ≥5)
    2. side effects remain acceptable
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.15 mg/kg/hour
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.2 mg/kg/hour
  * The maximum dose of ketamine will be limited to 300 mg per 24 hours
  The patient may receive ketamine up to 72 hours after initiation.
Arm/Group | Protocol for Administering Ketamine to Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Pain Scores of >2 Points on the Pain Scale
Description: Determine if there is an apparent improvement in pain control with the ketamine infusion based on the investigator's discretion and comparison to past pain scores. Pain was scored on a scale from 0 to 10. Zero equaled no pain and 10 equaled a lot of pain.
Time Frame: Baseline then daily while inpatient, up to 72 hours
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine: This group will receive ketamine
  ketamine: The medication will be administered intravenously. This study will utilize 4 doses of ketamine: 0.05 mg/kg/hour, 0.1 mg/kg/hour, 0.15 mg/kg/hour, and 0.2 mg/kg/hour.
  Dosing Regimen:
  * All patients will begin the ketamine infusion at 0.05 mg/kg/hour.
  * 4 or more hours after the infusion is started, the dose may be increased to 0.1 mg/kg/hour if:
    1. the patient's pain has not improved to an acceptable level (pain score is still ≥5)
    2. side effects remain acceptable
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.15 mg/kg/hour
  * 4 hours or more after the previous increase, the dose may be adjusted to 0.2 mg/kg/hour
  * The maximum dose of ketamine will be limited to 300 mg per 24 hours
  The patient may receive ketamine up to 72 hours after initiation.
Arm/Group | Ketamine
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Number of Participants Who Showed a Reduction of Opioid Utilization While on IV Ketamine
Description: Looking at the reduction of opioid utilization while on IV Ketamine. Three participants were enrolled in the study, therefore a comprehensive analysis could not be done due to the low enrollment.
Time Frame: Baseline then daily while inpatient, up to 72 hours
Measure: Count of Participants; unit: Participants
Groups:
- Ketamine: This group will receive ketamine
  ketamine: Medication administered via IV. This study will utilize 4 doses of ketamine: 0.05 mg/kg/hr, 0.1 mg/kg/hr, 0.15 mg/kg/hr, and 0.2 mg/kg/hr.
  Dosing Regimen:
  * Patients begin the ketamine infusion at 0.05 mg/kg/hr.
  * 4 or more hrs after infusion is started, the dose may be increased to 0.1 mg/kg/hr if:
    1. patient's pain has not improved to an acceptable level
    2. side effects remain acceptable
  * 4 hrs or more after the previous increase, the dose may be adjusted to 0.15 mg/kg/hr
  * 4 hrs or more after the previous increase, the dose may be adjusted to 0.2 mg/kg/hour
  * Maximum dose of ketamine is limited to 300 mg per 24 hrs
  Patient may receive ketamine up to 72 hrs after initiation.
Arm/Group | Ketamine
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Collected over 72 hour period
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No